CLINICAL TRIAL: NCT06108414
Title: The Efficacy and Safety of Low-dose Versus Standard-dose Rivaroxaban in Elderly Patients With Atrial Fibrillation
Brief Title: Low-dose Versus Standard-dose Rivaroxaban in Elderly Patients With Atrial Fibrillation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCRC2022002
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation; Anticoagulant Adverse Reaction; Stroke; Major Adverse Cardiac Events
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Cardiovascular Diseases | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose rivaroxaban (Experimental): 15mg q.d. rivaroxaban for 2 years after randomization. The dose should be reduced in the following special conditions: 1. Creatinine clearance <50 mL/min; 2. Body weight ≤60kg; 3. Age ≥80 years old. In the low-dose group, the dose was reduced from the usual 15mg q.d. to 10mg q.d. .
  Interventions: Drug: low-dose rivaroxaban
- Standard-dose rivaroxaban (Active Comparator): 20mg q.d. rivaroxaban for 2 years after randomization. The dose should be reduced in the following special conditions: 1. Creatinine clearance <50 mL/min; 2. Body weight ≤60kg; 3. Age ≥80 years old. In the standard-dose group, the dose was reduced from the 20mg q.d. to 15mg q.d. .
  Interventions: Drug: Standard-dose rivaroxaban

INTERVENTIONS:
Drug: low-dose rivaroxaban — Rivaroxaban 15mg q.d. (The dose should be reduced to 10mg q.d. in the following special populations: 1. Creatinine clearance <50 mL/min; 2. Body weight ≤60kg; 3. Age ≥80 years old)
  Arms: Low-dose rivaroxaban
Drug: Standard-dose rivaroxaban — Rivaroxaban 20mg q.d. (The dose should be reduced to 15mg q.d. in the following special populations: 1. Creatinine clearance <50 mL/min; 2. Body weight ≤60kg; 3. Age ≥80 years old)
  Arms: Standard-dose rivaroxaban

SUMMARY:
To evaluate the efficacy and safety of low-dose versus standard-dose rivaroxaban anticoagulation therapy in elderly patients with atrial fibrillation.

ELIGIBILITY:
Inclusion criteria:

* Age ≥70 years
* Patients with atrial fibrillation (atrial fibrillation rhythm of at least 30 seconds duration recorded by ECG or Holter within 1 year)
* CHA2DS2-VASc score ≥2 in men and ≥3 in women
* Able to cooperate in signing ICFs

Exclusion criteria：

* Moderate-to-severe mitral stenosis, or prior mechanical valve replacement surgery, or unresected atrial myxoma, or known left ventricular thrombus
* Prior biological valve replacement or valve repair surgery within 6 months
* Left ventricular assist device implantation status
* Severe stroke event within 3 months or any stroke within 14 days Major stroke events were defined as those with a Modified Rankin Scale score of 3-5.

Score 3: moderately disabled, requiring some assistance but walking without assistance; Score 4: severe disability, unable to walk independently, unable to meet their own needs without the help of others; Score 5: severe disability, bedridden, incontinent, requiring ongoing care and attention

* Transient ischemic attack (TIA) occurred within 3 days
* Transient atrial fibrillation due to reversible triggers (e.g., after cardiac surgery, pulmonary embolism, untreated hyperthyroidism)
* Prior or planning to undergo atrial fibrillation catheter ablation, drug cardioversion, electroconversion, or major surgery in 3 months; Prior catheter or surgical ablation > 3 months without atrial fibrillation electrocardiogram records
* Prior or planning to undergo left atrial appendage occlusion
* Active infective endocarditis
* High or increasing risk for bleeding i. Traumatic surgery that has been completed within the last 3 months or is planned within the next 3 months ii. Previous severe intracranial, intraocular, spinal cord, retroperitoneal, or nontraumatic intra-articular hemorrhage.

iii. Gastrointestinal bleeding within the past year iv. Symptomatic or gastroscopic peptic ulcer within the last month v. Hemorrhagic constitution or coagulopathy vi. Difficult-controlled hypertension (180mm Hg systolic and/or 100 mm Hg diastolic)

* Severe renal impairment (estimated creatinine clearance ≤ 15 mL/min)
* Active liver disease

Including but not limited to:

i. Persistent ALT, AST > 2×ULN; ii. TBil > 1.5×ULN; iii. Known active hepatitis A, B or C; iv. Cirrhosis

* Hemoglobin level <100g/L or thrombocytopenia count <100 × 10^9/L
* Having conditions warrant standard-dose or low-dose anticoagulation treatment (non-AF, such as VTE)
* Having conditions warrant warfarin anticoagulation treatment
* Daily dose of aspirin >100mg
* Having received dual antiplatelet therapy or intravenous antiplatelet drugs within 5 days (note: P2Y12 receptor antagonist alone or ≤ 100mg aspirin alone can be enrolled)
* Having received fibrinolysis treatment in 10 days or planning to use fibrinolytic drugs
* Having conditions warrant the following medications: CYP3A4 and P-gp inhibitors (itraconazole, ketoconazole, voriconazole, posaconazole, clarithromycin, erythromycin, fluconazole, ritonavir, dronedarone, etc.), selective serotonin reuptake inhibitors (SSRI)/serotonin norepinephrine reuptake inhibitors (SNRI) drugs (fluoxetine, paroxelin, etc.) CYP3A4 inducers (rifampicin, phenytoin, carbamazepine, phenobarbital, St. John's wort, etc.), long-term use of NSAIDs
* Having allergic or adverse reactions to any excipients (including but not limited to lactose, starch, etc.) in rivaroxaban tablets, including but not limited to hereditary lactose or galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, etc.
* Having diagnosed with malignant tumors within 6 months, or receiving radiotherapy/chemotherapy, with an expected lifespan of no more than 3 years
* Antiphospholipid syndrome
* Having been enrolled in another interventional clinical trial within the past 30 days or at the same time
* Mental disorders, communication barriers, cognitive impairment, or other serious illnesses that may affect the participation in this study
* Known poor adherence to study follow-up or taking study drugs
* Other conditions deemed by the investigator to be inappropriate for enrollment

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4374 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events(MACCE) | Through study completion, an estimated average of 2 years
  A composite endpoint of clinical events including cardiovascular death, myocardial infarction, stroke, and systemic embolism was firstly recorded after randomization

SECONDARY OUTCOMES:
Bleeding events | Through study completion, an estimated average of 2 years
  A composite endpoint of ISTH major bleeding events and clinically relevant non major bleeding events was recorded after randomization
Net clinical benefit | Through study completion, an estimated average of 2 years
  A composite endpoint of all-cause death, myocardial infarction, stroke, transient ischemic attack, systemic embolism, ISTH major bleeding events and clinically relevant non major bleeding events after randomization
Components of all primary and secondary outcome measures | Through study completion, an estimated average of 2 years
  All-cause death, myocardial infarction, stroke, transient ischemic attack, systemic embolism, ISTH major bleeding events and clinically relevant non major bleeding events after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- National Clinical Research Center for Cardiovascular Diseases, State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Han J, Qi W, Yuan S, Liu H, Wang Y, Zhang H, Liu J, Zhao Y, Zhang Y, Zheng L, Yao Y, Zheng Z. Efficacy and safety of low-dose rivaroxaban in elderly patients with atrial fibrillation for oral anticoagulation therapy: Rationale, design, and study protocol for a multicenter randomized controlled trial (SAFE-AF). Am Heart J. 2025 Dec;290:268-277. doi: 10.1016/j.ahj.2025.07.011. Epub 2025 Jul 15. PMID 40675206